CLINICAL TRIAL: NCT02625480
Title: A Phase 1/2 Multi-Center Study Evaluating the Safety and Efficacy of KTE-X19 in Pediatric and Adolescent Subjects With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia or Relapsed/Refractory B-Cell Non-Hodgkin Lymphoma (ZUMA-4)
Brief Title: Study Evaluating Brexucabtagene Autoleucel (KTE-X19) in Pediatric and Adolescent Participants With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia or Relapsed/Refractory B-Cell Non-Hodgkin Lymphoma
Acronym: ZUMA-4
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTE-C19-104; 2023-509440-97 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2015-12-05; First posted 2015-12-09 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia; Relapsed/Refractory B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell | interventions — brexucabtagene autoleucel; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by a single infusion of chimeric antigen receptor (CAR) transduced autologous T cells administered intravenously at a target dose of 2 x 10^6 anti-CD19 CAR+ T cells/kg or 1 x 10^6 anti-CD19 CAR+ T cells/kg.
  Interventions: Biological: Brexucabtagene Autoleucel (KTE-X19); Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Brexucabtagene Autoleucel (KTE-X19)
Drug: Fludarabine — Administered intravenously
Drug: Cyclophosphamide — Administered intravenously

SUMMARY:
The primary objectives of this study are to evaluate the safety and efficacy of brexucabtagene autoleucel (KTE-X19) in pediatric and adolescent participants with relapsed/refractory (r/r) B-precursor acute lymphoblastic leukemia (ALL) or relapsed or refractory (r/r) B-cell non-Hodgkin lymphoma (NHL).

As of October 2022, no further patients with acute B-cell Acute Lymphoblastic Leukemia (ALL) will be asked to join the study. The study remains open for recruitment for patients that have B-cell Non Hodgkin Lymphoma (NHL).

DETAILED DESCRIPTION:
All participants who received KTE-X19, and have completed at least 24 months of protocol assessments, will be transitioned to a separate long-term follow-up (LTFU) study. The purpose of the LTFU study (KT-US-982-5968.) is to complete the remainder of the 15-year follow-up assessments.

ELIGIBILITY:
Key Inclusion Criteria for the ALL Cohort

* Relapsed or refractory B-precursor ALL defined as one of the following:

  * Primary refractory disease
  * Any relapse within 18 months after first diagnosis
  * Relapsed or refractory disease after 2 or more lines of systemic therapy
  * Relapsed or refractory disease after allogeneic transplant provided individual is at least 100 days from stem cell transplant at the time of enrollment
* Disease burden defined as at least 1 of the following:

  * Morphological disease in the bone marrow (> 5% blasts)
  * Minimal/Measurable Residual Disease (MRD) positive (threshold 10^-4 by flow or Polymerase chain reaction (PCR))
* Individuals with Ph+ disease are eligible if they are intolerant to tyrosine kinase inhibitor (TKI) therapy, or if they have relapsed/refractory disease despite treatment with at least 2 different TKIs
* Age ≤ 21 years and weight ≥ 6 kg at the time of assent or consent per Institutional Review Board (IRB) guidelines
* Lansky (age < 16 years at the time of assent/consent) or Karnofsky (age ≥ 16 years at the time of assent/consent) performance status ≥ 80 at screening
* Adequate renal, hepatic, pulmonary and cardiac function defined as:

  * Creatinine clearance (as estimated by Cockcroft Gault or Schwartz) ≥ 60 mL/min
  * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 5 x upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 x ULN, except in individuals with Gilbert's syndrome
  * Left ventricular shortening fraction (LVSF) ≥ 30% or left ventricular ejection fraction (LVEF) ≥ 50%, as determined by an echocardiogram or multi-gated acquisition scan (MUGA), no evidence of pericardial effusion (except trace or physiological) as determined by an echocardiogram (ECHO) and no clinically significant arrhythmias
  * No clinically significant pleural effusion, pericardial effusion or ascites
  * Baseline oxygen saturation > 92% on room air

Key Exclusion Criteria for the ALL Cohort

* Diagnosis of Burkitt's leukemia/lymphoma according to the World Health Organization (WHO) classification or chronic myelogenous leukemia lymphoid blast crisis
* History of malignancy other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) unless disease free for at least 3 years
* History of severe hypersensitivity reaction to aminoglycosides or any of the agents used in this study
* Central nervous system (CNS) involvement and abnormalities:

  * Any CNS tumor mass by imaging and/or parameningeal mass (cranial and/or spinal)
  * Presence of central nervous system (CNS)-3 disease, defined as white blood cell (WBC) ≥ 5/µL in Cerebrospinal Fluid (CSF) with presence of lymphoblasts with or without neurologic symptoms
  * CNS-2 disease, defined as WBC < 5/µL in CSF with presence of lymphoblasts and with neurologic symptoms (see note below for further clarification).
  * Note: Neurologic symptoms may include but are not limited to cranial nerve palsy (if not explained by extracranial tumor) and clinical cord compression.
  * (Individuals with CNS-1 (no detectable lymphoblasts in the CSF) and those with CNS-2 without clinically evident neurological changes are eligible to participate in the study)
  * History or presence of CNS disorder, such as cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement, posterior reversible encephalopathy syndrome (PRES), or cerebral edema with confirmed structural defects not related to lymphoma by appropriate imaging. History of stroke or transient ischemic attack within 12 months before enrollment. Individuals with seizure disorders requiring active anticonvulsive medication.
* History of concomitant genetic syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman-Diamond syndrome or any other known bone marrow failure syndrome
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment
* History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months of enrollment.
* Primary immunodeficiency
* History of human immunodeficiency virus (HIV) infection or acute / chronic active hepatitis B or C infection. Individuals with a history of hepatitis infection must have cleared their infection as determined by standard serological and genetic testing per current Infectious Diseases Society of America guidelines or applicable country guidelines.
* Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management.
* Prior medication:

  * Prior CD19 directed therapy (other than blinatumomab), including CAR+ T cell, bispecific T cell engager (BiTE), and antibody drug conjugate (ADC), with the exception of individuals who received brexucabtagene autoleucel (KTE-X19) in this study and are eligible for re-treatment
  * Treatment with alemtuzumab within 6 months prior to leukapheresis, or treatment with clofarabine or cladribine within 3 months prior to leukapheresis
  * Donor lymphocyte infusion (DLI) within 28 days prior to enrollment
  * Any drug used for graft-versus-host disease (GVHD) within 4 weeks prior to enrollment
* Acute GVHD grade II-IV by Glucksberg criteria or severity B-D by IBMTR index; acute or chronic GVHD requiring systemic treatment within 4 weeks prior to enrollment
* Live vaccine ≤ 6 weeks prior to enrollment
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant. Females who have undergone surgical sterilization are not considered to be of childbearing potential
* Individuals of both genders of child-bearing potential who are not willing to use a birth control method considered to be highly effective per protocol from the time of consent through 6 months after conditioning chemotherapy or brexucabtagene autoleucel (KTE-X19) infusion, whichever is longer.

Key Inclusion Criteria for the NHL Cohort

* Histologically confirmed aggressive B cell NHL
* Relapsed or refractory histologically confirmed aggressive B-cell NHL per 1 or more of the following:

  * Primary refractory disease
  * Any relapse within 18 months after first diagnosis
  * Relapsed or refractory disease after 1 or more lines of systemic therapy
  * Relapsed or refractory disease after autologous /allogeneic stem cell transplant provided individual is at least 6 weeks from autologous stem cell transplant and at least 3 months from allogeneic stem cell transplant at the time of enrollment
* Individuals must have received adequate prior therapy including at a minimum all of the following:

  * Anti-CD20 monoclonal antibody, unless the investigator determines that the tumor is CD20 negative
  * An anthracycline-containing chemotherapy regimen
* Age <18 years old and weight ≥ 6kg
* Lansky (age < 16 years at the time of assent/consent) or Karnofsky (age ≥ 16 years at the time of assent/consent) performance status ≥ 80 at screening
* Adequate renal, hepatic, pulmonary, and cardiac function defined as the following:

  * Creatinine clearance (as estimated by Cockcroft Gault or Schwartz) ≥ 60 mL/min
  * Serum ALT/AST ≤ 5 ULN
  * Total bilirubin ≤1.5 x ULN except in individuals with Gilbert's syndrome
  * Left ventricular shortening fraction(LVSF) ≥ 30% or left ventricular ejection fraction (LVEF) ≥ 50%, as determined by ECHO or MUGA, no evidence of pericardial effusion (except trace or physiological) as determined by an ECHO, and no clinically significant arrhythmias
  * Baseline oxygen saturation > 92% on room air

Key Exclusion Criteria for the NHL Cohort

* History of malignancy other than nonmelanoma skin cancer, carcinoma in situ (eg, cervix, breast), or follicular lymphoma (FL) unless disease free for at least 3 years
* Autologous stem cell transplant within <6 weeks of planned KTE-X19 infusion; allogeneic stem cell transplant within <3 months of planned KTE-X19 infusion
* Prior CD19 targeted therapy other than blinatumomab and loncastuximab tesirine-lpyl
* History of severe, immediate hypersensitivity reaction attributed to aminoglycosides
* Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management.
* History of HIV infection or acute/chronic active hepatitis B or C infection. Individuals with a history of hepatitis infection must have cleared their infection as determined by standard serological and genetic testing per current Infectious Diseases Society of America guidelines or applicable country guidelines
* Acute GVHD grade II-IV by Glucksberg criteria or severity B-D by International Bone Marrow Transplant Registry (IBMTR) index; acute or chronic GVHD requiring systemic treatment within 4 weeks prior to enrollment.
* CNS involvement and abnormalities:

  * Any CNS tumor mass and/or parameningeal mass (cranial and/or spinal) by imaging with current or prior history of neurological symptoms within 3 months prior to screening.

Note: CNS involvement without neurologic symptoms will be allowed.

* History or presence of any CNS disorder such as a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, any autoimmune disease with CNS involvement, posterior reversible encephalopathy syndrome (PRES), or cerebral edema with confirmed structural defects by appropriate imaging. History of stroke or transient ischemic attack within 12 months before enrollment. Individuals with seizure disorders requiring active anti-convulsive medication.

  * History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment
  * Primary immunodeficiency
  * History of severe immediate hypersensitivity reaction to any of the agents used in this study
  * Live vaccine ≤ 6 weeks prior to planned start of lymphodepleting chemotherapy regimen
  * Individuals of both genders of child-bearing potential who are not willing to use a birth control considered to be highly effective per protocol from the time of consent through 12 months after the completion of lymphodepleting chemotherapy or brexucabtagene autoleucel (KTE-X19) infusion, whichever is longer.
  * Prior medication:
* Prior CD19 directed therapy (other than blinatumomab), including CAR+ T cell, BiTE, and ADC, with the exception of individuals who received brexucabtagene autoleucel (KTE-X19) in this study and are eligible for re-treatment
* Treatment with alemtuzumab within 6 months prior to leukapheresis, or treatment with clofarabine or cladribine within 3 months prior to leukapheresis
* DLI within 28 days prior to enrollment
* Any drug used for GVHD within 4 weeks prior to enrollment

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Percentage of Participants Experiencing Adverse Events Defined as Dose-Limiting Toxicities (DLT) | Up to 28 days
  Dose-limiting toxicity is defined as protocol-defined brexucabtagene autoleucel (KTE-X19)-related events with onset within the first 28 days following brexucabtagene autoleucel (KTE-X19) infusion.
Phase 2: Overall Complete Remission Rate in the ALL Cohort | Up to 24 months
  Overall complete remission rate will be determined per independent review.
Phase 2: Objective Response Rate in the NHL Cohorts | Up to 24 months
  Objective Response Rate will be determined per investigator review.

SECONDARY OUTCOMES:
Minimum Residual Disease Negative Remission Rate in the ALL Cohort | Up to 3 months
  Minimal residual disease (MRD) response rate is defined as MRD < 10^-4 per the standard assessment.
Allogeneic Stem Cell Transplant Rate in the ALL Cohort | Up to 24 months
  The incidence of allogeneic stem cell transplant will be analyzed.
Changes Over Time in Patient Reported Outcomes (PRO) Scores in the ALL and NHL Cohorts | Up to 10 years
  The PRO scores will be measured by the Pediatric Quality of Life Inventory (PedsQL) for children and adolescents and European Quality-of-Life-5 Dimension (EQ-5D) for all participants.
  The PedsQL comprises of 23 items in the dimensions of physical, emotional, social, and school functioning. Transformed total, physical health summary, and psychosocial health summary scores range from 0-100 with higher scores indicating better health-related quality of life.
  The EQ-5D is a generic questionnaire for assessing the participant's overall health status. The EQ-5D consists of a 5 dimension descriptive system including mobility, self-care, usual activities, pain/comfort, and anxiety/depression and a visual analogue scale (EQ-VAS) which allows the respondent to record health. The VAS allows a participant to indicate self-reported health on a vertical scale, ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). The PedsQL scores and EQ-5D scores will be reported.
Overall Complete Remission Rate in the ALL Cohort | Up to 10 years
Relapse-Free Survival for the ALL Cohort | Up to 24 months
  Relapse-Free Survival is defined as the time from the brexucabtagene autoleucel (KTE-X19) infusion date to the date of disease relapse or death from any cause.
Progression Free Survival in the NHL Cohort | Up to 10 years
Overall Survival in the ALL and NHL Cohorts | Up to 10 years
  Overall survival is defined as the time from brexucabtagene autoleucel (KTE-X19) infusion to the date of death from any cause.
Duration of Remission in the ALL and NHL Cohorts | Up to 24 months
  Duration of remission is defined as the time between the participant's first complete response per independent review to relapse or any death in the absence of documented relapse.
Percentage of Participants with Anti-Brexucabtagene Autoleucel (KTE-X19) Antibodies in Blood in the ALL and NHL Cohorts | Up to 10 years
Percentage of Participants Experiencing Adverse Events and Common Terminology Criteria for Adverse Events (CTCAE) Grade Changes in Safety Laboratory Values in ALL and NHL Cohorts | Up to 10 years
CR Rate Within 3 Months Per Independent Review in ALL Cohorts | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (30):
- United States (15):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - University of Miami Hospital & Clinics, Miami, Florida
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Columbia University Irving Medical Center/Morgan Stanley Children's Hospital-NYP, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Monroe-Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - University of Virginia Health System, Pediatric Hematology/Oncology Clinic, Charlottesville, Virginia
- University Hospital Gent, Ghent, Belgium
- The Hospital for Sick Children, Toronto, Canada
- University Hospital Brno, Brno, Czechia
- France (4):
  - Unité d'Oncologie et Hématologie Pédiatriques, Bordeaux
  - Institut d'Hematologie et Oncologie Pediatrique, Lyon
  - Hopital d'Enfants la Timone, Marseille
  - Hopital Robert Debre - Sevice d'Hemato-immunologic, Paris
- University Medical Center Hamburg-Eppendorf (UKE), Hamburg, Germany
- Bambino Gesù Children's Hospital, Rome, Italy
- Prinses Maxima Centrum, Utrecht, Netherlands
- Poland (2):
  - Jurasz University Hospital 1; Collegium Medicum, Bydgoszcz
  - Wroclaw Medical University, Wroclaw
- Spain (2):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitario La Paz, Madrid
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wayne AS, Huynh V, Hijiya N, Rouce RH, Brown PA, Krueger J, Kitko CL, Ziga ED, Hermiston ML, Richards MK, Baruchel A, Schuberth PC, Rossi J, Zhou L, Goyal L, Jain R, Vezan R, Masouleh BK, Lee DW. Three-year results from phase I of ZUMA-4: KTE-X19 in pediatric relapsed/refractory acute lymphoblastic leukemia. Haematologica. 2023 Mar 1;108(3):747-760. doi: 10.3324/haematol.2022.280678. PMID 36263840
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KTE-C19-104